CLINICAL TRIAL: NCT01407159
Title: ASSIST - A Study in SurvIvors of Type B Aortic Dissection Undergoing Stenting
Brief Title: A Study in SurvIvors of Type B Aortic Dissection Undergoing Stenting
Acronym: ASSIST
Status: Completed | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ASSIST
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Type B Aortic Dissection
Keywords: type b dissection; thoracic stentgraft; aortic stent; clinical and technical success; safety and feasibility of E-XL aortic stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Thoracic Stentgraft plus E-XL: male and female patients with complicated type B aortic dissection involving the infra-diaphragmatic aorta treated with any thoracic stentgraft extended by the E-XL aortic stent
- Control group: historical control group fulfilling the following criteria:
  * Age +/- 3 years
  * Sex matched
  * Same follow-up period

SUMMARY:
Cohort study according to national regulatory guidelines: Non-interventional, observational cohort study. Pair-matched comparison with patients chosen from historical series.

To evaluate the clinical and technical success as well as the safety and feasibility of the E-XL aortic stent used in complicated type B aortic dissection in addition to a classic stentgraft in a single procedure.

ELIGIBILITY:
The clinical records of the patients mus support the following criteria:

* Age > 18 years
* Type B dissection with expanding false lumen eligible for endovascular treatment which occured within 90 days prior to implantation
* The endovascular treatment may be associated with a complementary surgical operation
* The total diameter of the dissected aortic segment should not surpass 6cm, and have increased between 0.5 and 1cm within 1 month, prior to implantation
* Visceral arteries involvement, i.e. perfusion of side branches via true or false lumen of type B dissection
* Aortic kinking < 90°
* The patient must be available for the appropriate follow-up times for the duration of the study
* Informed consent from patient or authorized relative

The data of whose patients clinical records confirm one of the following conditions will not be considered in this study:

* Patients with a contraindication as indicated in the instruction for use
* Patients with chronic thrombocytopenia or ongoing anticoagulation
* Patients with renal failure and/or creatinine >2.4mg/dl immediately before the intervention
* Patients in whom the false lumen is completely thrombosed
* Patients with ongoing infection
* Patients with ongoing cancer
* Patients who are enrolled in a clinical study
* Aortic landing zone diameter over 40 mm
* Potentially emboligenic iliac and aortic atheroma lesions
* Associated pathology with life expectancy of less than 24 months
* Unstable infectious syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with complicated type B aortic dissection involving the infra-diaphragmatic aorta
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical and technical success as well as the safety and feasibility of the E-XL aortic stent used in complicated type B aortic dissection in addition to a classic thoracic stent-graft in a single procedure. | February 2014

CONTACTS AND LOCATIONS:
Locations (15):
- Germany (9):
  - Klinikum Augsburg, Augsburg
  - German Heart Center, Berlin
  - University Hospital, Essen
  - University Hospital, Freiburg im Breisgau
  - Hannover Medical School, Hanover
  - University Hospital, Jena
  - University Hospital Munich Grosshadern, Munich
  - St. Franziskus Hospital, Münster
  - University Hospital, Rostock
- Italy (2):
  - Department of Radiologia Toracica e Vascolare, Bologna
  - IRCCS Policlinico San Donato Milano, Milan
- Poland (2):
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
- Spain (2):
  - Thorax Insitute, Hospital Clinic, University of Barcelona, Barcelona
  - Hospital Clinico Universitario de Valladolid, Valladolid

REFERENCES:
- [Derived] Nienaber CA, Yuan X, Aboukoura M, Blanke P, Jakob R, Janosi RA, Lovato L, Riambau V, Trebacz J, Trimarchi S, Zipfel B, van den Berg JC; ASSIST study group. Improved Remodeling With TEVAR and Distal Bare-Metal Stent in Acute Complicated Type B Dissection. Ann Thorac Surg. 2020 Nov;110(5):1572-1579. doi: 10.1016/j.athoracsur.2020.02.029. Epub 2020 Mar 20. PMID 32205112